CLINICAL TRIAL: NCT02009007
Title: Effect of Phenylephrine or Dopamine Infusion on Cerebral Oxygen Saturation in Thoracic Surgery Patients
Brief Title: Vasopressors for Cerebral Oxygenation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-09-058
Record Dates: First submitted 2013-11-13; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Hypoxia; Hypotension
Keywords: cerebral oximeter; one lung ventilation; dopamine; phenylephrine
MeSH Terms: conditions — Hypoxia; Hypotension | interventions — Dopamine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dopamine (Experimental): dopamine is administered to maintain systolic blood pressure in the range of 80-120% of baseline during operation
  Interventions: Drug: dopamine
- phenylephrine (Experimental): Phenylephrine is administered to maintain systolic blood pressure in the range of 80-120% of baseline during operation
  Interventions: Drug: phenylephrine

INTERVENTIONS:
Drug: dopamine — continuous infusion during operation
  Arms: dopamine
Drug: phenylephrine — continuous infusion of phenylephrine during operation
  Arms: phenylephrine

SUMMARY:
Liberal fluid administration is one of risk factors of developing acute lung injury (ALI) in thoracic surgery. Therefore, the investigators try to restrain fluid administration, and in the case of intraoperative hypotension, the investigators often administer vasoactive agents or inotropes. One lung ventilation (OLV) which is routinely employed for thoracic surgery decrease arterial oxygenation and oxygen delivery to brain can be also decreased. In this study, the investigators compared dopamine and phenylephrine in respect to maintaining cerebral oxygen saturation in major thoracic surgery. The investigators hypothesis is that dopamine is better than phenylephrine to maintain cerebral oxygen saturation in thoracic surgery.

DETAILED DESCRIPTION:
A 'restrictive' intraoperative fluid regimen, avoiding hypovolaemia but limiting infusion to the minimum necessary reduced major complications after complex surgery. This restrictive fluid regimen is especially relevant in thoracic surgery since acute lung injury is known to be related to large amount of fluid administration during operation to treat hypotension. One study suggests that, for every 500-mL increase in perioperative fluids, there is an odds ratio of 1.17 for developing ALI after lung resection. Slinger suggested that fluid should be restricted just to the point of maintaining urine output of 0.5 mL/kg/h, and vasopressors may be used if tissue perfusion is inadequate. Therefore, restriction of fluid administration and treatment of hypotension which is not caused by major hemorrhage with vasoactive agents could be a basic concept in thoracic anesthesia.

Patients who undergoing lung resection surgery usually receive one lung ventilation (OLV). Decrease of systemic oxygenation occurs during OLV due to intrapulmonary shunt. During OLV, significant decrease in cerebral oxygenation (SctO2) is also known to occur and low SctO2 is related to postoperative complications.

Because the endpoint of hemodynamic optimization is to improve oxygen delivery to major organs, understanding how the administration of vasoactive agents affects cerebral perfusion and oxygenation, the most important organ in the body is of major clinical relevance. Recently published studies show that near-infrared spectroscopy (NIRS)-guided brain protection protocols might lead to reduced neurocognitive complications and improved postoperative outcomes.

However, there have been no data on which agent between dopamine and phenylephrine, the most commonly used aged during operation against hypotension, is better in maintaining cerebral oxygen saturation during thoracic surgery. Therefore, the investigators try to compare dopamine and phenylephrine continuous infusion in respect to maintaining SctO2 in major thoracic surgery.

In addition, acute kidney injury (AKI) develops in around 6% of patients after lung resection surgery and AKI is related to poor prognosis and prolonged duration of hospital admission.Therefore, the investigators also tried to find which agent is better to maintain urinary output during operation and reduce postoperative AKI. The investigators also found there is difference in postoperative delirium incidence between dopamine and phenylephrine continuous infusion.

The primary aims of the study were (i) to investigate the effect of phenylephrine and dopamine continuous infusion on cerebral SctO2 (ii) to identify the hemodynamic variables [mean blood pressure, cardiac output, heart rate (HR), stroke volume (SV)] which are responsible for the changes in cerebral SctO2 induced by phenylephrine and dopamine treatments.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* American society of anesthesia physical status I-III

Exclusion Criteria:

* Symptomatic cardiovascular disease
* Poorly controlled hypertension (systolic arterial pressure ≥160 mm Hg)
* Cerebrovascular disease
* Poorly controlled diabetes mellitus (blood glucose ≥200 mg/dl)
* Diuretics or antidepressant use before operation
* Renal insufficiency (creatinine>1.5 mg/dl)
* Cerebral infarction
* Documented coagulopathy

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral oximeter reading | at 60 minutes after one lung ventilation

SECONDARY OUTCOMES:
cardiac output | at 60 minutes after one lung ventilation
incidence of delirium | participants will be followed for the first 48 hours of ICU stay
incidence of acute renal injury | participants will be followed for the first 48 hours of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea